CLINICAL TRIAL: NCT05739162
Title: Endoscopic Sleeve Gastroplasty (ESG) as a Treatment Option for Obesity in Ulcerative Colitis (UC) Patients Undergoing Colectomy With Ileal Pouch Anal Anastomosis (IPAA)
Brief Title: A Study of Endoscopic Sleeve Gastroplasty for Obesity in Ulcerative Colitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Amanda M. Johnson, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-007643
Record Dates: First submitted 2023-02-13; First posted 2023-02-22 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Obesity; Ulcerative Colitis
Keywords: ESG; IPAA
MeSH Terms: conditions — Obesity; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Endoscopic Sleeve Gastroplasty (ESG) (Experimental): Participants undergo Endoscopic Sleeve Gastroplasty (ESG). Following the 6-week transitional diet after undergoing the ESG procedure, participants will start the lifestyle intervention.
  Interventions: Device: Apollo Endoscopic Suture System; Behavioral: Lifestyle Intervention

INTERVENTIONS:
Device: Apollo Endoscopic Suture System — Endoscopic Sleeve Gastroplasty (ESG), and endoscopic minimally-invasive weight loss procedure, utilizing a suturing device to reduce the stomach volume by 70-80% through the creation of sleeve. This is accomplished by a series of endoscopically placed stitches through the stomach wall.
Behavioral: Lifestyle Intervention — Low-calorie healthy diet personalized by a dietician according to individual patients' needs and conducive to weight loss. Physical activity will be encourage and assessed.

SUMMARY:
The purpose of this research is to gather information on the safety and effectiveness of Endoscopic Sleeve Gastroplasty (ESG) for weight loss in a population of obese UC patients undergoing colectomy with eventual IPAA.

ELIGIBILITY:
Inclusion Criteria:

* BMI 30-50 kg/m2 for at least 6 months prior to ESG
* Diagnosis of UC with plans to undergo or who have already undergone colectomy as part of a plan to pursue eventual 3-stage ileal pouch anal anastomosis (IPAA)
* Willing to adhere to the diet and behavior modifications required for ESG
* Able to follow the visit schedule
* Able to provide informed consent
* If female, be either post-menopausal, surgically sterile, or agree to practice birth control during year of study and have negative serum Human Chorionic Gonadotropin (HCG) at screening/baseline

Exclusion Criteria:

* Prior gastric or bariatric surgery or other alteration to upper gastrointestinal anatomy which would preclude safe or technical performance of ESG
* Current or recent (last six months) gastric or duodenal ulceration
* Esophageal or gastric varices
* Significant motility disorder of the esophagus or stomach
* Large hiatal hernia measuring >5 cm or ≤ 5 cm and associated with severe gastroesophageal reflux
* Severe coagulopathy, hepatic insufficiency, or cirrhosis
* Gastric mass
* Presence of any other medical condition which precludes safe performance of elective endoscopy such as poor general health and/or history of severe hepatic, cardiac, or pulmonary disease
* Serious or uncontrolled psychiatric illness which may compromise patient understanding of procedure or compliance with follow-up visits
* Unwilling to participate in an established diet and behavior modification program, with routine follow-up
* Ongoing corticosteroid use at a dose of >5 mg daily
* Daily use of anti-inflammatory agents such as non-steroidal medications, or anticoagulants without medical supervision
* Alcohol or drug addiction
* Females who are pregnant, nursing, or planning pregnancy within the next year
* Concomitant use of or unwillingness to avoid any use of weight loss medications, weight loss supplements, or weight loss herbal preparations
* Has a condition or is in a situation which in the investigator's opinion may put the subject at significant risk or may interfere significantly with the subject's participation in the study

Ages: 22 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Percent total body weight loss | 6 months
  Percent total body weight loss (%TBWL) calculated by the equation ((baseline screening weight in kilograms (kg) subtracted by follow-up weight in kg) divided by baseline screening weight in kg) times 100.
Number of subjects with serious adverse events | 24 months
  Total number of subjects to report serious adverse event related to the ESG procedure

SECONDARY OUTCOMES:
Number of early peri-operative complications | 1 year following procedure
  Number of early (less than 30 days) peri-operative complications related to IPAA and ileostomy takedown clinical standard of care procedure
Number of late peri-operative complications | 1 year following procedure
  Number of late (greater than 30 days) peri-operative complications related to IPAA and ileostomy takedown clinical standard of care procedure
Change gastrointestinal symptom rating scale (GSRS) | Week 4, Week 12, Week 24, 12 months post-ileostomy takedown
  ESG tolerance measured by GSRS which includes 15 items and utilizes a 7-point response scale to measure a participant's level of discomfort associated with a given GI symptom, ranging from "No discomfort at all" to "Very severe discomfort."
Modified pouchitis disease activity index (mPDAI) | 12 months post-ileostomy takedown
  Assess overall pouch function one year following ileostomy takedown using the modified pouchitis disease activity index (mPDAI) score. The mPDAI quantitates clinical symptoms and endoscopic features (edema, granularity, friability, loss of vascular pattern, mucus exudate, and ulceration) on several separate 0-2 point scores, whereby a total score greater than or equal to 5 is indicative of pouchitis.
Durable weight loss | 12 months and 12 months post-ileostomy takedown
  Number of subjects to achieve durable weight loss

CONTACTS AND LOCATIONS:
Overall Officials: Amanda M Johnson, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/cls-20556627